CLINICAL TRIAL: NCT05480566
Title: Effects of Functional Strength Training and Neuromuscular Electrical Stimulation During Hospitalisation for Acute Exacerbation of Chronic Obstructive Pulmonary Disease: a Randomised Controlled Trial
Brief Title: Functional Strength Training and Neuromuscular Electrical Stimulation in Severe Acute Exacerbations of COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The anticipated intervention could not be delivered due to low admission time
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Chris Burtin, Assistant Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOF20BL20
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Acute Exacerbation of COPD
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; Inpatient; Functional strength training; NMES
MeSH Terms: interventions — Oxygen; Methylprednisolone; fenoterol, ipratropium drug combination; Dosage Forms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional strength training + NMES (Experimental): The experimental group will receive the standard of care plus functional strength training and quadriceps neuromuscular electrical stimulation. Functional strength training will include lower limb (e.g. rising from chair, heel rises) and upper limb (e.g. push-ups from the chair and against the wall) exercises for 15 min/day. Target levels of dyspnoea and/or perceived exertion will be 4 to 6 in the modified Borg scale. For neuromuscular electrical stimulation, electrodes will be placed longitudinally on the vastus intermedius and vastus medialis and a symmetric biphasic pulse waveform, with a pulse duration of 400ms, a frequency of 50Hz, in cycles of 8s of contraction and 20s of rest, will be used for 30min/day. The highest intensity tolerated by the patient will be used and intensity will be increased every time the patient feels comfortable with increasing the intensity. The device Compex Pro Rehab (CE-0473) will be used.
  Interventions: Other: Functional strength training; Device: NMES; Drug: Daily medical treatment (e.g., oxygen, medrol, duovent, azitromycine); Other: Routine physiotherapy
- Standard of care (Active Comparator): The standard of care group will receive the common treatment delivered at the hospital, i.e., routine medical treatment and daily sessions of approximately 15 minutes consisting of airway clearance techniques and breathing exercises upon indication, mobilization, and low-intensity daily walking/cycling exercise (5 to 10 minutes) according to patients' tolerance.
  Interventions: Drug: Daily medical treatment (e.g., oxygen, medrol, duovent, azitromycine); Other: Routine physiotherapy

INTERVENTIONS:
Other: Functional strength training — Functional strength training will include lower limb (e.g. rising from chair, heel rises) and upper limb (e.g. push-ups from the chair and against the wall) exercises for 15 min/day. Target levels of dyspnoea and/or perceived exertion will be 4 to 6 in the modified Borg scale.
  Arms: Functional strength training + NMES
Device: NMES — For neuromuscular electrical stimulation, electrodes will be placed longitudinally on the vastus intermedius and vastus medialis and a symmetric biphasic pulse waveform, with a pulse duration of 400ms, a frequency of 50Hz, in cycles of 8s of contraction and 20s of rest, will be used for 30min/day. The highest intensity tolerated by the patient will be used and intensity will be increased every time the patient feels comfortable with increasing the intensity. The device Compex Pro Rehab (CE-0473) will be used.
  Arms: Functional strength training + NMES
Drug: Daily medical treatment (e.g., oxygen, medrol, duovent, azitromycine) — Patients will be treated with daily medication prescribed by the physician, which can include oxygen, medrol, duovent, azitromycine or other medications that physicians consider that are needed.
  Other Names: Medication
Other: Routine physiotherapy — Daily sessions of approximately 15 minutes consisting of airway clearance techniques and breathing exercises upon indication, mobilization, and low-intensity daily walking/cycling exercise (5 to 10 minutes) according to patients' tolerance.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is highly prevalent and frequently punctuated by severe acute exacerbations (AECOPD), defined as a temporary worsening of symptoms which leads to hospitalisation. AECOPD result in physical inactivity, muscle weakness and decreased exercise capacity, which impacts negatively on patients' health status, and increases patients' susceptibility for new exacerbations and death. To date, light aerobic exercises, such as early mobilisation and low-intensity ambulation, have become part of standard of care during severe AECOPD. Nevertheless, additional strength training using neuromuscular electrical stimulation and functional exercises, which have been shown to prevent skeletal muscle dysfunction whilst inducing minimal stress in the ventilatory system, might be of added value to optimize patients' functional performance and symptoms during activities at discharge.

Therefore, this randomized controlled trial aims to evaluate the effectiveness of additional functional strength training and neuromuscular electrical stimulation on top of standard of care during hospitalisation for an AECOPD to enhance functional performance, symptoms of dyspnoea and fatigue during activities, and readmission rate.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive and life-threatening condition characterised by persistent respiratory symptoms and airflow limitation. It affects 384 million people, is one of the main causes of morbidity and the third cause of mortality worldwide, responsible for around 3 million deaths annually. Consequently, COPD results in significant and increasing health, economic and social burden. The trajectory of COPD is frequently punctuated by acute exacerbations (AECOPD), defined as episodes of acute worsening of respiratory symptoms that result in additional therapy.

Severe AECOPD lead to hospitalization and account for more than 70% of all COPD-related costs. AECOPD are associated with physical inactivity, quadriceps muscle weakness and decreased exercise capacity, which impacts negatively on patients' health status, and increases patients' susceptibility for exacerbations recurrence, hospitalisations and death. Therefore, minimising the negative sequelae of AECOPD and preventing rehospitalisation are fundamental treatment goals for individuals, families and health, economic and social systems.

People discharged from the hospital after an AECOPD benefit from participating in pulmonary rehabilitation, but uptake is generally low. By all means, however, it is important to maximize the patient's functional performance and minimize symptoms during activities by the time of discharge. During an AECOPD, patients experience increased dyspnoea. Consequently, exercise modalities with minimal ventilatory requirements are preferred. To date, light aerobic exercises, such as early mobilisation and low-intensity ambulation, have become part of the standard of care. Nevertheless, additional strength training using neuromuscular electrical stimulation (NMES) and functional exercises, which have been shown to prevent skeletal muscle dysfunction whilst inducing minimal stress in the ventilatory system, might be of added value to optimize patients' functional performance and symptoms at discharge.

The researchers hypothesise that adding functional strength training and NMES to the standard mobilisation practice during hospitalisation for an AECOPD will: i) preserve or enhance patients' functional performance; ii) reduce symptoms of dyspnoea and fatigue and iii) decrease the short-term readmission rate.

Therefore, this study aims to evaluate the impact of adding functional strength training and NMES to standard mobilisation practice during hospitalisation for an AECOPD on:

* functional performance (primary outcome);
* symptoms of dyspnoea and fatigue (secondary outcome);
* readmission rate (exploratory outcome).

Hospitalised patients with AECOPD will be recruited consecutively at the hospital "Ziekenhuis Oost-Limburg" (ZOL). Patients will be eligible if they are: i) hospitalised due to an AECOPD according to the Global Initiative for Chronic Obstructive Lung Disease criteria, ii) included within 48h of hospital admission and iii) able to provide informed consent. Exclusion criteria will include: i) need for mechanical ventilation or admission in the intensive care unit; ii) unstable cardiovascular disease; iii) hospitalization in the previous month; iv) significant musculoskeletal or neuromuscular impairment that precludes the performance of the tests or participation in the study; v) signs of cognitive impairment; vi) current neoplastic or immunological disease; vii) implantable electronic devices (e.g., pacemaker, implantable cardioverter defibrillator (ICD), cardiac resynchronization therapy (CRT) device) and viii) sensitivity alterations.

A randomised controlled trial will be conducted. Researchers will provide patients with a brief explanation about the study, clarify any doubts and collect the informed consent. Patients will be assessed at 3 timepoints: within 48h of hospital admission (baseline assessment), at the day of discharge (post assessment) and 1 month after discharge (1-month follow-up). Additionally, patients' clinical records will be checked to assess for new AECOPD-related hospitalisations up to 6 months after discharge.

After baseline assessment, patients will be randomly allocated (ratio 1:1) to either the experimental or standard of care group. Randomisation will be performed using a random number generator. Both groups will receive daily treatment until discharge. All treatment sessions will be performed by the experienced physiotherapist team in the hospital and/or by a trained member of the research team not involved in the assessments. Patients' symptoms, vital signs and peripheral oxygen saturations will be monitored in all sessions.

The standard of care group will receive the common treatment delivered at the hospital, i.e., routine medical treatment and daily sessions of approximately 15 minutes consisting of airway clearance techniques and breathing exercises upon indication, mobilization, and low-intensity daily walking/cycling exercise (5 to 10 minutes) according to patients' tolerance.

The experimental group will receive the standard of care plus functional strength training and quadriceps neuromuscular electrical stimulation. Functional strength training will include lower limb (e.g. rising from chair, heel rises) and upper limb (e.g. push-ups from the chair and against the wall) exercises for 15 min/day. Target levels of dyspnoea and/or perceived exertion will be 4 to 6 in the modified Borg scale. For NMES, electrodes will be placed longitudinally on the vastus intermedius and vastus medialis and a symmetric biphasic pulse waveform, with a pulse duration of 400ms, a frequency of 50Hz, in cycles of 8s of contraction and 20s of rest, will be used for 30min/day. The highest intensity tolerated by the patient will be used and intensity will be increased every time the patient feels comfortable with increasing the intensity. The device "Compex Pro Rehab" (CE-0473) will be used.

All the assessments will be performed by an experienced physiotherapist, blinded to the allocation group. All the measurements will be done at the hospital "Ziekenhuis Oost-Limburg".

Sociodemographic, anthropometric (i.e., height and weight to compute body mass index) and general clinical data, as well as prior spirometric measurement, will be collected from clinical records for patients' characterization. Functional performance (the primary outcome) will be measured with the 1-minute sit-to-stand test. Isometric quadriceps strength and handgrip strength will be assessed at right and left sides. Self-reported symptoms, functional status and impact of the disease will also be collected (modified British Medical Research Council dyspnoea questionnaire, Functional Assessment of Chronic Illness Therapy-Fatigue, London chest activities of daily living, COPD Assessment Test). Physical activity will be objectively quantified, as an exploratory outcome, with an Actigraph GT3X. Additionally, the number of new AECOPD-related hospitalisations up to 6 months after discharge will be retrieved from clinical records.

A sample size estimation based on preliminary data from an exploratory study was performed to detect a moderate effect size (f=0.2), with 80% power, 5% significance level and moderate correlation among repeated measure (r=0.5) on the 1-minute sit-to-stand test. Considering that in rehabilitation interventions during hospitalization drop-out rates are around 6% (25, 26), 30 patients with AECOPD per group will be needed.

Descriptive statistics (i.e., mean and standard deviation, median and interquartile range, and/or relative percentages) will be used to describe the sample. Data collected at the 3 timepoints will be compared between the standard of care and intervention groups using inferential statistics. Normality of the data distribution will be explored with histograms, Q-Q plots and Shapiro-Wilk or Kolmogorov-Smirnov tests. Independent t-tests for normally distributed data and Mann Whitney U-tests for ordinal and non-normally distributed data will be used to compare baseline measurements between the 2 groups. Chi-square or Fisher's Exact tests will be used for categorical data. Comparisons between groups and timepoints will be performed using a two-way mixed ANOVA for normally distributed data, or the Kruskal-Wallis test with Bonferroni-adjusted pairwise comparisons for the non-normally distributed data. All statistical analysis will be performed in the software Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* hospitalised due to an AECOPD according to the Global Initiative for Chronic Obstructive Lung Disease criteria
* included within 48h of hospital admission
* able to provide informed consent
* dutch speaker

Exclusion Criteria:

* need for mechanical ventilation or admission in the intensive care unit
* unstable cardiovascular disease
* hospitalization in the previous month
* significant musculoskeletal or neuromuscular impairment that precludes the performance of the tests or participation in the study
* signs of cognitive impairment
* current neoplastic or immunological disease
* implantable electronic devices (e.g., pacemaker, implantable cardioverter defibrillator [ICD], cardiac resynchronization therapy [CRT] device)
* sensitivity alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
1-minute sit-to-stand test | within 48 hours of hospital admission (baseline assessment)
  Functional performance (the primary outcome) will be measured with the 1-minute sit-to-stand test, which is a valid, reliable and responsive test to assess this outcome in patients with chronic obstructive pulmonary disease (COPD). A straight-backed armless chair of 46-48 centimeters, with a hard seat, stabilized against a wall will be used to perform the test. Participants will be asked to sit with their hands stationary on the hips, without using the hands or arms to assist movement and instructed to stand up all the way and sit down, as many times as possible, in 1 minute. The protocol described by Crook et al will be followed. Since this test presents no learning effect, only one measurement will be asked in each timepoint.
Change in the 1-minute sit-to-stand test | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  Functional performance (the primary outcome) will be measured with the 1-minute sit-to-stand test, which is a valid, reliable and responsive test to assess this outcome in patients with chronic obstructive pulmonary disease (COPD). A straight-backed armless chair of 46-48 centimeters, with a hard seat, stabilized against a wall will be used to perform the test. Participants will be asked to sit with their hands stationary on the hips, without using the hands or arms to assist movement and instructed to stand up all the way and sit down, as many times as possible, in 1 minute. The protocol described by Crook et al will be followed. Since this test presents no learning effect, only one measurement will be asked in each timepoint.

SECONDARY OUTCOMES:
Change in Isometric quadriceps strength | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  A hand-held dynamometer (Microfet, Biometrics, NL) will be used to assess right and left isometric quadriceps strength, which has shown good test-retest reliability. Patients will be seated with the knee and hip flexed at 90º. With the dynamometer positioned stable proximal to the ankle, on the anterior surface of the leg, the assessor will apply resistance and instruct the patients to perform a maximal contraction against the resistance (make test). Three repetitions will be performed on each side and the highest value will be used for analysis.
Change in Handgrip strength | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  Right and left handgrip strength will be assessed isometrically using a hand-held dynamometer (Jamar, Preston, MI, USA). Patients will be seated with the elbow of the arm holding the dynamometer flexed at 90º and touching the side of the chest, and the forearm and wrist in neutral position. Three maximal efforts will be performed on each side and the best will be used for analysis.
Change in the modified British Medical Research Council dyspnoea questionnaire (mMRC) | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  The modified British Medical Research Council dyspnoea questionnaire (mMRC) is a simple, valid and widely used instrument to characterise the impact of dyspnoea on the daily activities of patients with chronic obstructive pulmonary disease (COPD). mMRC comprises five grades (statements) in a scale from 0 to 4, with higher grades indicating greater perceived respiratory limitation.
Change in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is a valid and reliable multidimensional questionnaire to assess tiredness, weakness, and difficulty in handling daily activities due to fatigue in patients with chronic obstructive pulmonary disease (COPD). The FACIT-F includes 13-item, each item has a 5-points Likert scale (from "not at all" to "very much"), and scores range from 0 to 52, with higher scores indicating less fatigue.
Change in the London chest activities of daily living questionnaire (LCADL) | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  Self-reported functional status will be assessed with the London chest activities of daily living questionnaire (LCADL), a valid tool designed to assess activities of daily living in patients with COPD. LCADL comprises 15 questions divided into four domains. Each question is scored on a 0-5 scale, with 5 representing the greatest dyspnea-related impairment in activities of daily living. The total score can range from 0 to 75 points, with higher scores indicating greater limitation in activities of daily living.
Change in the COPD Assessment Test (CAT) | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment, usually up to 7 days after admission), 1 month after hospital discharge (1-month follow-up)
  Impact of the disease will be measured with the disease-specific questionnaire COPD Assessment Test (CAT), which is a valid and reliable instrument for use in patients with AECOPD. CAT consists of eight items (i.e., cough, sputum, chest tightness, breathlessness going up hills/stairs, activity limitations at home, confidence leaving home, sleep and energy) scored from 0 to 5. The individual score of each item is added to provide a total score that can range from 0 to 40, with higher scores indicating higher impact of the disease.
Number of new exacerbation-related hospitalisations | 6 months after hospital discharge
  The number of new exacerbation-related hospitalisations up to 6 months after discharge will be retrieved from clinical records.

OTHER OUTCOMES:
Change in Daily physical activity | During hospitalization (i.e., from hospital admission until hospital discharge), at 1-month follow-up (i.e., 1-month after hospital discharge)
  Physical activity will be objectively quantified, as an exploratory outcome, with an Actigraph GT3X (Actigraph LLC Pensacola, FL, USA). The ActiGraph GT3X is a small, lightweight three-axial accelerometer (3.8x3.7x1.8 cm) with a sample frequency of 30Hz, which provides activity data in a scale from 0 to 15,000 counts/min. Data will be processed with ActiLife software version 5.10.0. The monitor will be worn at the waist level using a comfortable elastic strap. Patients will wear the monitor during hospitalization and for 7 consecutive days at 1-month follow-up. Patients will be asked to wear the device continuously, except during bathing/showering and sleeping. Days with less than 8 hours of wearing time will be excluded from the analysis. Patients will not be included in the analysis if they did not have at least 3 valid weekdays of measurement.
Change in Body mass index | within 48 hours of hospital admission (baseline assessment), 1 month after hospital discharge (1-month follow-up)
  Patients' body mass index will be computed in kg/m^2 based on patients' height and weight.
Change in Heart rate | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment), 1 month after hospital discharge (1-month follow-up)
  Heart rate will be assessed in beats per minute using a oximeter and blood pressure meter. It will be assessed in the different study timepoints and, in addition, to ensure patients' safety through the intervention sessions, heart rate will be monitored in every intervention session.
Change in Respiratory rate | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment), 1 month after hospital discharge (1-month follow-up)
  Respiratory rate will be assessed by direct observation, counting the number of respiratory cycles.
Change in Blood pressure | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment), 1 month after hospital discharge (1-month follow-up)
  Blood pressure (both systolic blood pressure and diastolic blood pressure) will be assessed using a blood pressure meter.
Peripheral oxygen saturation | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment), 1 month after hospital discharge (1-month follow-up)
  Peripheral oxygen saturation will be assessed with a pulse oximeter. It will be assessed in the different study timepoints and, in addition, to ensure patients' safety through the intervention sessions, peripheral oxygen saturation will be monitored in every intervention session.
modified Borg scale | within 48 hours of hospital admission (baseline assessment), at the day of hospital discharge (post assessment), 1 month after hospital discharge (1-month follow-up)
  Patients' self-reported level of dyspnea and fatigue will be collected at rest, using the modified Borg scale. In addition, these levels will be collected after the different exercises to monitor the exercise intensity. The modified Borg scale ranges from 0 to 10 with higher scores indicating higher perceived dyspnea/fatigue symptoms.
Change in Lung function | within 48 hours of hospital admission (baseline assessment), 1 month after discharge (1-month follow-up)
  Prior spirometric measurement will be collected from clinical records to assess the forced expiratory volume in 1 second and, therefore, the degree of bronchial obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Burtin, PhD, Principal Investigator — Rehabilitation Research Center (REVAL), Faculty of Rehabilitation Sciences, Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No